CLINICAL TRIAL: NCT05144321
Title: Constitution of a Prospective Twin Pregnancy Cohort in Order to Study the Risk Factors for Obstetric Complications COGEM
Brief Title: Twin Pregnancy Cohort
Acronym: COGEM
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0703
Record Dates: First submitted 2021-11-24; First posted 2021-12-03 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Pregnant With Complication; Twin Pregnancy With Antenatal Problem
Keywords: Pregnant women; Environment; Adverse outcome; Age >18 years; Gestational age >25 weeks; Delivery of a twin pregnancy
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All pregnant women delivering a twin pregnancy: All pregnant women delivering a twin pregnancy
  Interventions: Other: Impact of environment upon obstetrical; Other: neonatal and maternal adverse outcome

INTERVENTIONS:
Other: Impact of environment upon obstetrical — Impact of environment upon obstetrical
Other: neonatal and maternal adverse outcome — neonatal and maternal adverse outcome

SUMMARY:
The investigators know that multiple factors are involved in the risk of obstetric complications. The twin pregnancy model appears to be an interesting model for a bio-statistical analysis of data collected in the context of a complete pregnancy, in particular because it can reveal differences for a common exposure.

The aim of the study is to constitute a prospective cohort of twin pregnancies. The collection of data on the health of mothers, pregnancies, childbirth, and the health of twins at birth should make it possible to reveal results with sufficient statistical power for a prospective study.

ELIGIBILITY:
Inclusion criteria:

* Pregnant women
* Delivery of a twin pregnancy
* Gestational age >25 weeks
* Age >18 years

Exclusion criteria:

* Singleton pregnancy
* Miscarriage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women delivering a twin pregnancy
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
maternal adverse outcome | day 1
  Pomaternal adverse outcome

SECONDARY OUTCOMES:
Neonatal adverse outcome | day 1
  Neonatal adverse outcome
Obstetrical adverse outcome | day 1
  Obstetrical adverse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC